CLINICAL TRIAL: NCT06621550
Title: The Effect of High-Intensity Interval Training Exercise on Cognitive Function of Young Adults: A Pilot Randomized Controlled Trial
Brief Title: Effect of High-Intensity Interval Training Exercise on Cognitive Function of Young Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Freddy Man Hin LAM, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20231129004
Record Dates: First submitted 2024-09-29; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Young Healthy Adults
Keywords: Executive Functions; High Intensity Interval Training; Young Healthy Adults
MeSH Terms: interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIIT Arm (Experimental): Participants will receive a single session of HIIT, which lasts for 19 minutes
  Interventions: Other: High Intensity Interval Training
- Control Arm (No Intervention): Participants will be arranged to rest quietly on a chair for 19 minutes.

INTERVENTIONS:
Other: High Intensity Interval Training — Participants will receive a single session of HIIT, which last for 19 minutes in duration. During the HIIT session, participants will complete 2 minutes stretching warm-up exercise, followed by a video of exercises which will be projected on the screen to facilitate the participants to follow. The exercise in the video involves various combinations of aerobic and core resistance exercise such as squat jump, jump lunge, push up, burpee, mountain climber etc. The exercise involved bodyweight or minimal basic equipment only, the workout to rest ratio is 45 secs: 15 secs. Participants' heart rate will be kept surveillance and to maintain their respective heart rate attained 85% of aged predicted maximal heart rate during the workout period.
  Arms: HIIT Arm

SUMMARY:
To explore the sustainability of the acute effect of High Intensity Interval Training (HIIT) on executive function in young adults.

ELIGIBILITY:
Inclusion Criteria:

* Young adult aged 18-40 years old
* No visionary defect or other sensory condition including uncorrected refractive defect and color blindness refraining the individual to be assessed by the tasks

Exclusion Criteria:

* With known neurological, cardiovascular, or other physical and mental conditions that limit the ability to safely participate in high-intensity interval training
* With known specific learning disabilities
* Known drug or alcohol abuse problems

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Stroop task | From baseline to 72 hours post intervention
  Stroop Task is a neurocognitive test for the performance on inhibition control. Participants are shown a series of word colors that are either congruent or incongruent with the color of the word itself. The participant is required to respond to the color of the word and not the word itself.

SECONDARY OUTCOMES:
Flanker Task | From baseline to 72 hours post intervention
  Flanker Task is a neurocognitive test for the performance on inhibition control. Participants are shown a series of arrows. The participant is to respond to which way the center arrow is pointing; whether it is to the right or to the left
Trail making test (TMT) | From baseline to 72 hours post intervention
  TMT is a neurocognitive test for the performance on cognitive flexibility. There are part A and part B in the TMT. The time required to completed part A as well as part B would be recorded separately, the difference in time in completing part B and part A (B-A) and the ratio of time in completing part A and part B (B/A) would be used as the interference score.
Wisconsin Card Sorting test (WCST) | From baseline to 72 hours post intervention
  WCST is a neurocognitive test for the performance on cognitive flexibility. Participants will be presented with four response cards, which are of different geometric properties (number of objects, color of object and shape of objects), and one stimulus card at a time. Participants will be required to sort the stimulus card. There are 30 trials in the test, number of correct sorting will be recorded, and accuracy will be obtained as number of correct sorting divided by 30.
Change in accuracy as measured by the 2-back task | From baseline to 72 hours post intervention
  2-back task is a neurocognitive test for the performance on working memory. Participants are presented with a sequence of stimuli in character form. The task consists of indicating when the current stimulus matches the one from 2 steps earlier in the sequence. There are 48 trials in the task, the number of correct responses will be recorded. The accuracy will be obtained as number of correct responses divided by 39.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hung Hom, Hong Kong

IPD SHARING:
Plan to Share IPD: No